CLINICAL TRIAL: NCT02378532
Title: A Phase I Trial for the Addition of Chloroquine, an Autophagy Inhibitor, to Concurrent Chemoradiation for Newly Diagnosed Glioblastoma
Brief Title: The Addition of Chloroquine to Chemoradiation for Glioblastoma
Acronym: CHLOROBRAIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLOROBRAIN
Record Dates: First submitted 2015-02-12; First posted 2015-03-04 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Glioblastoma Multiforme
Keywords: Glioblastoma; Chloroquine; Autophagy; EGFRvIII; Radiotherapy; Temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Chloroquine; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy/Temozolomide + Chloroquine (Experimental): Eligible patients will receive radiotherapy and chemotherapy according to standard protocol for newly diagnosed GBM.
  Chloroquine will be escalated in 3 dose-levels (200mg, 400mg and 600mg) up each containing a minimum of 3 and a maximum of 6 patients. Based on the results of the DSMB, an additional level of 300mg was added.
  Interventions: Drug: Chloroquine; Radiation: Radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Chloroquine — Three cohorts of 3 patients will receive chloroquine in escalating doses (3 dose levels: 200 mg up to 600 mg daily) during standard treatment (radiotherapy and temozolomide) for newly diagnosed GBM. Extra patients can be added to a cohort in case of dose limiting toxicity, resulting in a maximum of 6 patients per dose level. Based on the results of the DSMB an additional leven of 300mg was added.
Radiation: Radiotherapy — Patients will receive megavoltage radiotherapy in a conventionally fractionated regimen of 59.4 Gy in 33 fractions in 6.5 weeks, using modern computer-based treatment planning and delivery techniques. Treatment should start within 6 weeks of surgery.
Drug: Temozolomide — Patients will take TMZ 75 mg/m² po qd during the course of radiotherapy six adjuvant cycles of TMZ. After a 4 week break, patients will receive up to six cycles of adjuvant oral TMZ 150 - 200 mg/m² po qd for 5 days every 28 days. The starting dose is 150 mg/m² po qd. At the start of cycle 2 the dose will be escalated to 200mg/m2, if the CTC non-hematologic toxicity for cycle 1 is grade ≤2 (except for alopecia, nausea, and vomiting), absolute neutrophil count is ≥1.5 x 109/L and the platelet count ≥ 100 x 109/L.
  Other Names: Temodal

SUMMARY:
Patients with a glioblastoma (GBM) have a poor prognosis with a median survival of 14.6 months after maximal treatment with a resection and chemoradiation. Since the pivotal trial evaluating the effect of temozolomide (TMZ), overall survival has not increased.

Treatment of GBM xenografts in vivo with chloroquine (CQ), an antimalarial agent, has been shown to reduce the hypoxic fraction and sensitizes tumors to radiation. Epidermal growth factor receptor (EGFR) amplification or mutation is regularly observed GBM and is thought to be a major contributor to radioresistance. The most common EGFR mutation in GBM (EGFRvIII) is present in 50-60% of patients whose tumor shows amplification of EGFR. EGFR provides cells with a survival advantage through autophagy when exposed to stresses such as hypoxia and nutrient starvation. This effect is even more pronounced in EGFRvIII overexpressing tumors. Previously, the potential effect CQ has been demonstrated in a small randomized controlled trial in GBM treated with radiotherapy and carmustine, which showed a trend towards increased overall survival. However, as the intracellular effects of chloroquine are dose-dependent the maximum tolerated dose for CQ in combination with concurrent radiotherapy with daily temozolomide needs to be established.

DETAILED DESCRIPTION:
This trial has been designed as an open label, single center combination phase I trial. The primary objective is to determine the maximum tolerated dose (MTD) for chloroquine (CQ) in combination with concurrent radiotherapy with daily temozolomide in patients with a newly diagnosed GBM.

Eligible patients will receive radiotherapy and chemotherapy according to standard protocol for newly diagnosed GBM. This consists of 33 daily fractions of 1.8 Gy to the tumor and surrounding margin in combination with TMZ 75 mg/m² per os daily (po qd) and six adjuvant cycles of TMZ 150 - 200 mg/m² po qd. Treatment will be combined with daily intake of escalating doses of chloroquine. Chloroquine will start with week before the start of radiotherapy and end on the last day of radiotherapy.

The rate of subject entry and escalation to the next dose level will depend upon assessment of the safety profile of patients entered at the previous dose level. Toxicity will be evaluated according to the NCI common Terminology Criteria for Adverse Events (CTCAE), Version 4.0.

The 3 + 3 cohort method is used. A minimum of three patients will be entered at each dose level. All three will be followed during the concomitant radiotherapy and a 4 week observation period before escalation to the next dose level.

The start dose is 200mg chloroquine daily. Before opening the next higher dose level all toxic effects at the preceding dose level will be reviewed and expansion or escalation will be undertaken as appropriate

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade IV supratentorial astrocytoma (glioblastoma multiforme)
* Tumor tissue available for histopathological analysis (MGMT, EGFRvIII)
* Diagnosis must have been made by biopsy or resection ≤ 3 months prior to study entry
* 18 years or older
* Karnofsky performance status ≥ 70
* Absolute neutrophil count at least 1.5 x 109/L and platelets at least 100 x109/L
* Adequate renal function
* Adequate hepatic function
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Females must have negative results for pregnancy tests performed
* No breast feeding.
* If male, subject must be surgically sterile or practicing a method of contraception

Exclusion Criteria:

* Prior radiotherapy
* Prior chemotherapy
* Recent (< 3 months) severe cardiac disease (NYHA class >1) (congestive heart failure, infarction)
* History of cardiac arrythmia (multifocal premature ventricular contractions, uncontrolled atrial fibrillation, bigeminy, trigeminy, ventricular tachycardia) which is symptomatic and requiring treatment (CTC AE 4.0), or asymptomatic sustained ventricular tachycardia. Asymptomatic atrial fibrillation controlled on medication is allowed.
* Cardiac conduction disturbances or medication potentially causing them
* Treatment with investigational drugs in 4 weeks prior to or during this study
* If the subject has clinically significant and uncontrolled major medical condition(s) including but not limited to:

  * uncontrolled nausea/vomiting/diarrhea:
  * active uncontrolled infection, including HIV and hepatitis (HBV, HCV)
  * psychiatric illness/social situation that would limit compliance with study requirements
  * any medical condition, with the opinion of the study investigator, places the subject at an unacceptably high risk for toxicities.
* The subject has had another active malignancy within the past 3 years except for any cancer in situ that the principal Investigator considers to be cured.
* Chronic systemic immune therapy (with the exception of corticosteroids)
* Concurrent cytochrome P450 enzyme-inducing anticonvulsant drugs (e.g., phenytoin, carbamazepine, phenobarbital, primidone, or oxcarbazepine)
* Known glucose-6-phosphate dehydrogenase deficiency
* Psoriasis or porphyria
* Known hypersensitivity to 4-aminoquinoline compound
* Retinal or visual field changes unrelated to the tumor location prior to 4-aminoquinoline compound use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Toxicity (CTC AE 4.0 | up to 2.5 years
  Determining the MTD of chloroquine as a radiosensitizer

SECONDARY OUTCOMES:
Pharmacokinetics of chloroquine, desethylchloroquine, bisdesethylchloroquine. Profile parameters will include trough level (Cmin), AUC and elimination half-life. | up to 2 years
  Pharmacokinetic sampling will be done at the start of week 1 and week 2 to determine the interpatient variability and steady state and at the end of radiotherapy/TMZ/CQ and before the start of adjuvant temozolomide in order to determine the time to eliminate CQ from the body.
Presence of autophagic markers (LC3 and autophagic vesicles) | up to 2 years
  Evaluation of autophagic markers will be done at baseline, 2 weeks and at the end of chloroquine treatment
Evaluation of EGFRvIII status in histopathological material | up to 2 years
  During biopsy or tumor resection, a small piece of tissue will be collected to evaluate EGFRvIII status

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, prof., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- Maastricht Radiation Oncology, Maastricht, Netherlands

REFERENCES:
- [Background] Jutten B, Rouschop KM. EGFR signaling and autophagy dependence for growth, survival, and therapy resistance. Cell Cycle. 2014;13(1):42-51. doi: 10.4161/cc.27518. Epub 2013 Dec 13. PMID 24335351
- [Background] Rouschop KM, van den Beucken T, Dubois L, Niessen H, Bussink J, Savelkouls K, Keulers T, Mujcic H, Landuyt W, Voncken JW, Lambin P, van der Kogel AJ, Koritzinsky M, Wouters BG. The unfolded protein response protects human tumor cells during hypoxia through regulation of the autophagy genes MAP1LC3B and ATG5. J Clin Invest. 2010 Jan;120(1):127-41. doi: 10.1172/JCI40027. Epub 2009 Dec 14. PMID 20038797
- [Result] Sotelo J, Briceno E, Lopez-Gonzalez MA. Adding chloroquine to conventional treatment for glioblastoma multiforme: a randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2006 Mar 7;144(5):337-43. doi: 10.7326/0003-4819-144-5-200603070-00008. PMID 16520474
- [Result] Jutten B, Keulers TG, Schaaf MB, Savelkouls K, Theys J, Span PN, Vooijs MA, Bussink J, Rouschop KM. EGFR overexpressing cells and tumors are dependent on autophagy for growth and survival. Radiother Oncol. 2013 Sep;108(3):479-83. doi: 10.1016/j.radonc.2013.06.033. Epub 2013 Jul 25. PMID 23891088